CLINICAL TRIAL: NCT00684567
Title: SCH 52365 Phase II Clinical Study in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Temozolomide Phase II Clinical Study in Patients With Newly Diagnosed Glioblastoma Multiforme (Study P04661)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04661; JPC-05-351-22
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2009-03-12 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): It is the only arm of the study. Subjects receive a combination of radiotherapy and temozolomide, and then temozolomide monotherapy.
  Interventions: Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy will be administered in combination with temozolomide during the concomitant radiotherapy phase. Radiotherapy will consist of a conventionally fractioned regimen, delivering a total dose of 60 Gy in 6 weeks, in a once daily schedule of 2 Gy per fraction, for a total of 30 fractions. Radiation will be provided by a linear accelerator of x ray energy of 4 MV or higher.
  Other Names: Irradiation, radiation therapy
Drug: Temozolomide — During the concomitant radiotherapy phase (6 weeks), temozolomide will be administered in combination with radiotherapy, once daily at 75 mg/m2/day. Then, during the monotherapy phase, subjects will receive 6 cycles of temozolomide alone. Each cycle will last 28 days, and temozolomide will be administered once daily from Day 1 to Day 5 of each cycle. The dose of temozolomide in the first cycle will be 150 mg/m2/day, and may be increased to 200 mg/m2/day for Cycle 2 and subsequent cycles depending on nonhematologic toxicity observed and neutrophil and platelet count values. Capsules containing 5 mg, 20 mg, or 100 mg of temozolomide will be combined to achieve each subject's calculated dose.
  Other Names: Temodal, Temodar, SCH 052365

SUMMARY:
The purpose of this study is to evaluate the safety of combination therapy of radiotherapy and temozolomide ("concomitant radiotherapy phase"), and then temozolomide monotherapy ("monotherapy phase"), in patients with newly diagnosed glioblastoma multiforme. Progression free survival and response rate will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed newly diagnosed glioblastoma multiforme with WHO grade IV.
* Histological diagnosis must be made locally after biopsy or neurosurgical tumor resection.
* Four or more unstained tissue sections or a paraffin block must be provided to the Pathological Judgment Committee as tissue specimens.
* Initial surgery/biopsy at diagnosis performed <=6 weeks (42 days) prior to treatment with temozolomide.
* Age: >=18 and <=70 years.
* ECOG performance status <=2.
* Stable, non-increasing dose of corticosteroids over the 14 days prior to treatment with temozolomide.
* No prior chemotherapy or radiotherapy.
* Laboratory test values obtained within 14 days before initiation of administration of temozolomide must satisfy the following criteria:

  * absolute neutrophil count >= 1500/mm^3;
  * platelet count >= 100,000/mm^3;
  * serum creatinine <=1.5 times the upper limit of laboratory normal;
  * total bilirubin <=1.5 times the upper limit of laboratory normal;
  * glutamic oxaloacetic transaminase or glutamic pyruvic transaminase <2.5 times the upper limit of laboratory normal;
  * alkaline phosphatase < 2.5 times the upper limit of laboratory normal.
* Absence of pathological conditions that interfere with taking oral drugs.
* Contraception during the study period (from informed consent to the day of the last observation/examination of this study) is required in sexually active, potentially fertile patients, regardless of sex, under the supervision of the investigator or sub-investigator.
* The investigator and/or subinvestigator must judge that life expectancy is 12 weeks or more.
* Patients may be included regardless of sex or inpatient/outpatient.

Exclusion Criteria:

* Extensively disseminated glioblastoma multiforme.
* Severe disorders in the heart, liver, kidney, blood, etc.
* Presence of previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and non melanoma skin cancer.
* Women who are pregnant or lactating.
* Women who may be pregnant or who could become pregnant and do not adopt contraception method(s).
* Participation in another clinical study within 6 weeks prior to the initiation of administration of temozolomide.
* Subjects who the investigator and/or subinvestigator judged inappropriate to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09-27 (Actual); Primary Completion 2007-10-31 (Actual); Study Completion 2007-10-31 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiotherapy/Temozolomide: It is the only arm of the study. Subjects receive a combination of radiotherapy and temozolomide, and then temozolomide monotherapy.
Period: Concomitant Radiotherapy Period
Arm/Group | Radiotherapy/Temozolomide
Started | 30
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 2
Period: Monotherapy Period
Arm/Group | Radiotherapy/Temozolomide
Started | 23 (5 subjects completed radiotherapy combined therapy phase but did not proceed to monotherapy phase.)
Completed | 9
Not Completed | 14
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Progression of primary disease | 11

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy/Temozolomide
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Centralized Pathologic Diagnosis [Number; unit: Participants]
  High Grade Astrocytoma | 1
  Glioblastoma Multiforme | 27
  Anaplastic Astrocytoma | 1
  Gliosarcoma | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — 6-point, ordinal scale specifying patient's ability to perform activities from 0 (fully active) to 5 (dead).
  Participants
    0 | 14
    1 | 11
    2 | 5
    3 | 0
    4 | 0
    5 | 0
Type of Surgery [Number; unit: Participants]
  Radical Extraction | 7
  Partial Extraction | 21
  Biopsy | 2

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events With an Incidence of Greater Than or Equal to 20%
Description: Safety was assessed from the start of administration during the concomitant radiotherapy phase until 30 days after the completion of administration of monotherapy. Adverse events were classified under the system organ class using MedDRA-J Version 11.0.
Time Frame: until 30 days after the completion of administration of monotherapy
Measure: Number; unit: Participants
Arm/Group | Radiotherapy/Temozolomide
Number analyzed (Participants) | 30
Participants
  alopecia | 25
  nausea | 17
  anorexia | 17
  constipation | 15
  malaise | 14
  rash | 11
  weight decreased | 11
  headache | 10
  vomiting | 9
  dry skin | 8
  nasopharyngitis | 8
  diarrhea | 7
  convulsion | 7
  pruritus | 6
  neutrophil count decreased | 6
  wound complication | 6

2. Primary Outcome: Adverse Drug Reactions With an Incidence of Greater Than or Equal to 20%
Description: Safety was assessed from the start of administration during the concomitant radiotherapy phase until 30 days after the completion of administration of monotherapy.
Time Frame: until 30 days after the completion of administration of monotherapy
Measure: Number; unit: Participants
Arm/Group | Radiotherapy/Temozolomide
Number analyzed (Participants) | 30
Participants
  constipation | 15
  nausea | 11
  vomiting | 6
  neutrophil count decreased | 6
  weight decreased | 6
  malaise | 7
  anorexia | 9

3. Primary Outcome: Abnormal Changes in Laboratory Test Values With an Incidence of Greater Than or Equal to 20%
Description: as for outcome 2
Time Frame: until 30 days after the completion of administration of monotherapy
Measure: Number; unit: Participants
Arm/Group | Radiotherapy/Temozolomide
Number analyzed (Participants) | 30
Participants
  lymphocyte count decreased | 24
  white blood cell count decreased | 14
  eosinophil percentage increased | 10

4. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) for 1 Year
Description: Administration of SCH 52365 was continued until progression was observed (progression was judged by the investigator based on MRI and clinical symptoms).
Time Frame: 1 year after the start of admininstration in the concomitant radiotherapy phase
Measure: Number; unit: Participants
Arm/Group | Radiotherapy/Temozolomide
Number analyzed (Participants) | 30
Participants | 11 [20.1 to 53.4]

5. Secondary Outcome: Number of Participants With a Response (Complete Response [CR] + Partial Response [PR]) in Terms of Overall Tumor Response
Description: CR = measurable lesion disappeared.
  PR = total sum of lesions measurable in bidimension decreased by 50% or more on whole and no secondary progression attributable to tumor was noted. No onset of new lesion.
Time Frame: 1 year after the start of administration in the concomitant radiotherapy phase
Population: Response rate in terms of tumor response (ratio of CR + PR) in 19 participants was assessed by Efficacy and Safety Evaluation Committee. 19 participants were found to have measurable lesions. Nineteen participants (as opposed to 30 participants) were analyzed because that is how many participants were still alive 1 year after start of therapy.
Measure: Number; unit: Participants
Arm/Group | Radiotherapy/Temozolomide
Number analyzed (Participants) | 19
Participants | 6 [12.6 to 56.6]

ADVERSE EVENTS:
Arm/Group | Radiotherapy/Temozolomide
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy/Temozolomide (N=30)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
NECROSIS (General disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 2 (2)
EPILEPSY (Nervous system disorders) | 2 (3)
HYDROCEPHALUS (Nervous system disorders) | 1 (1)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (1)
PARALYSIS (Nervous system disorders) | 1 (1)
TONIC CONVULSION (Nervous system disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy/Temozolomide (N=30)
EAR DISCOMFORT (Ear and labyrinth disorders) | 3 (3)
EYE PAIN (Eye disorders) | 2 (2)
VISUAL DISTURBANCE (Eye disorders) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 15 (19)
DIARRHOEA (Gastrointestinal disorders) | 7 (12)
GASTRITIS (Gastrointestinal disorders) | 3 (3)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 17 (21)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 5 (7)
STOMATITIS (Gastrointestinal disorders) | 2 (3)
VOMITING (Gastrointestinal disorders) | 9 (17)
FATIGUE (General disorders) | 2 (3)
INFLAMMATION OF WOUND (General disorders) | 3 (3)
MALAISE (General disorders) | 14 (23)
PYREXIA (General disorders) | 5 (7)
NASOPHARYNGITIS (Infections and infestations) | 8 (9)
OTITIS EXTERNA (Infections and infestations) | 4 (4)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 5 (5)
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 2 (2)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 6 (7)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3)
BASOPHIL PERCENTAGE INCREASED (Investigations) | 2 (2)
BLOOD ALBUMIN DECREASED (Investigations) | 3 (3)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (7)
BLOOD CHLORIDE DECREASED (Investigations) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 4 (4)
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 3 (4)
BLOOD UREA INCREASED (Investigations) | 4 (5)
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 (2)
EOSINOPHIL PERCENTAGE INCREASED (Investigations) | 10 (16)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 25 (43)
MONOCYTE PERCENTAGE INCREASED (Investigations) | 2 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 7 (12)
PLATELET COUNT DECREASED (Investigations) | 4 (4)
PROTEIN TOTAL DECREASED (Investigations) | 4 (4)
WEIGHT DECREASED (Investigations) | 11 (15)
WEIGHT INCREASED (Investigations) | 4 (4)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 14 (28)
ANOREXIA (Metabolism and nutrition disorders) | 17 (28)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
CONVULSION (Nervous system disorders) | 6 (11)
DIZZINESS (Nervous system disorders) | 3 (3)
DYSKINESIA (Nervous system disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 10 (18)
HEMIPLEGIA (Nervous system disorders) | 3 (3)
HYPOAESTHESIA (Nervous system disorders) | 3 (4)
MEMORY IMPAIRMENT (Nervous system disorders) | 2 (2)
SENSORY DISTURBANCE (Nervous system disorders) | 3 (3)
SOMNOLENCE (Nervous system disorders) | 2 (2)
TREMOR (Nervous system disorders) | 3 (3)
INSOMNIA (Psychiatric disorders) | 4 (6)
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 25 (25)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 8 (10)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (7)
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (7)
RASH (Skin and subcutaneous tissue disorders) | 11 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No